CLINICAL TRIAL: NCT00217126
Title: Long-term Kidney Function (2 Arms-Prospective and Retrospective)
Brief Title: The Study of Long-term Deterioration of Kidney Transplants.
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Hennepin County Medical Center, Minneapolis (Other); University of Alabama at Birmingham (Other); University of Alberta (Other); University of Iowa (Other)
Responsible Party: Dr. Fernando Cosio, Mayo Clinic
Other Study IDs: 143-05
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is being done to create a kidney transplant database with information from many transplant centers for the purpose of studying ways to help improve transplant outcomes and the care of transplant recipients. This is also being done to learn why kidney transplant recipients have worsening of their kidney function, and whether there are specific findings that could result in future treatments.

DETAILED DESCRIPTION:
Data will be collected from the participant's medical records, local health care providers and participant's to clarify or add any information. Participants will have samples of blood, and urine obtained during their routine visits, that will be saved for testing in this study. In addition, participant's receiving a kidney biopsy performed as a part of their clinical care, will have a piece of the biopsy used for the study. This study will be followed for five years.

ELIGIBILITY:
In the prospective group, all participants who will be receiving a kidney transplant are eligible. In the retrospective group, kidney transplant recipients who are undergoing a kidney biopsy to determine the cause of change in their serum creatine level.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Kidney Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 870 (Actual)
Dates: Start 2005-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando G. Cosio, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States